CLINICAL TRIAL: NCT01536886
Title: A Phase 2 Study Comparing Treatment With LEO 90100 With Calcipotriol Plus Betamethasone Ointment, LEO 90100 Vehicle and Ointment Vehicle in Subjects With Psoriasis Vulgaris.
Brief Title: LEO 90100 Compared With Calcipotriol Plus Betamethasone Dipropionate Ointment, LEO 90100 Vehicle and Ointment Vehicle in Subjects With Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LEO 90100-35
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2016-08

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Betamethasone; calcipotriene; Ointments

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- LEO 90100 vehicle (Placebo Comparator): Aerosol foam with no active ingredient
  Interventions: Drug: LEO 90100 vehicle
- Betamethasone plus calcipotriol (Active Comparator): Calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate) ointment
  Interventions: Drug: Betamethasone plus calcipotriol
- LEO 90100 (Experimental): LEO 90100 aerosol foam: calcipotriol 50 mcg/g and betamethasone 0.5 mg/g (as dipropionate)
  Interventions: Drug: LEO 90100
- Ointment vehicle (Placebo Comparator): Ointment with no active ingredients
  Interventions: Drug: Ointment vehicle

INTERVENTIONS:
Drug: LEO 90100
  Arms: LEO 90100
Drug: Betamethasone plus calcipotriol
  Arms: Betamethasone plus calcipotriol
Drug: Ointment vehicle
  Arms: Ointment vehicle
Drug: LEO 90100 vehicle
  Arms: LEO 90100 vehicle

SUMMARY:
The purpose of this study is to investigate whether LEO 90100 and calcipotriol plus betamethasone are effective in the treatment of psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained prior to any trial related activities (including washout period).
* Age 18 years or above
* Either sex
* Any race or ethnicity
* All skin types
* Females of childbearing potential must have a negative pregnancy test at Day 0 (Visit 1).
* Females of childbearing potential must agree to use a highly effective method of birth control during the study. A highly effective method of birth control is defined as one which results in a low failure rate (less than 1% per year).
* Able to communicate with the investigator and understand and comply with the requirements of the study.

Exclusion Criteria:

* Systemic treatment with biological therapies, whether marketed or not, with a possible effect on psoriasis vulgaris within the following time periods prior to randomisation:

  * etanercept - within 4 weeks prior to randomisation
  * adalimumab, alefacept, infliximab - within 8 weeks prior to randomisation
  * ustekinumab - within 16 weeks prior to randomisation
  * other products - 4 weeks/5 half-lives (whichever is longer)
* Systemic treatment with all other therapies with a possible effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, methotrexate, ciclosporin and other immunosuppressants) within 4 weeks prior to randomisation.
* Subjects who have received treatment with any nonmarketed drug substance (i.e. a drug which has not yet been made available for clinical use following registration) within 4 weeks/5 half-lives (whichever is longer) prior to randomisation.
* PUVA therapy within 4 weeks prior to randomisation.
* UVB therapy within 2 weeks prior to randomisation.
* Planned excessive exposure of area(s) to be treated with study medication to either natural or artificial sunlight (including tanning booths, sun lamps, etc.) during the study.
* Planned initiation of, or changes to, concomitant medication that could affect psoriasis vulgaris (e.g. beta blockers, antimalarial drugs, lithium, ACE inhibitors) during the study.
* Current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis.
* Subjects with any of the following conditions present on the treatment area: viral (e.g. herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, icthyosis, ulcers and wounds.
* Other inflammatory skin disorders (e.g. seborrhoeic dermatitis or contact dermatitis) on the treatment area that may confound the evaluation of psoriasis vulgaris.
* Known or suspected disorders of calcium metabolism associated with hypercalcaemia.
* Known or suspected severe renal insufficiency or severe hepatic disorders.
* Known or suspected hypersensitivity to component(s) of the investigational products.
* Current participation in any other interventional clinical study.
* Previously randomised in this study.
* Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koo, MD, Principal Investigator — University of California, San Francisco School of Medicine
Locations (39):
- United States (39):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Dermatology Research Associates, Los Angeles, California
  - Dermatology Specialists, Inc., Oceanside, California
  - Skin Surgery Medical Group, Inc, San Diego, California
  - University Clinical Trials, Inc., San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - About Skin Dermatology and DermSurgery, PC, Denver, Colorado
  - Colorado Medical Research Center, Inc, Denver, Colorado
  - Horizons Clinical Research Center, Denver, Colorado
  - Dermatology Associates and Research, Coral Gables, Florida
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Gwinnett Clinical Research Ctr, Inc, Snellville, Georgia
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Glazer Dermatology, Buffalo Grove, Illinois
  - Clinical Research Advantage, Inc./Hudson Dermatology, LLC, Evansville, Indiana
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Owensboro Dermatology Associates, Owensboro, Kentucky
  - David Fivenson, MD, PLC, Ann Arbor, Michigan
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Derm Center, Troy, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Psoriasis Treatment Center of Central NJ, East Windsor, New Jersey
  - The Dermatology Group, PC, Verona, New Jersey
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Derm Research Center of New York, Stony Brook, New York
  - Philadelphia Institute of Dermatology, Fort Washington, Pennsylvania
  - Menter Dermatology Research Institute, Dallas, Texas
  - Suzanne Bruce and Associates, P.A.,The Center for Skin Research, Houston, Texas
  - Center for Clinical Studies, Houston, Texas
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koo J, Tyring S, Werschler WP, Bruce S, Olesen M, Villumsen J, Bagel J. Superior efficacy of the fixed combination calcipotriene plus betamethasone dipropionate in a novel aerosol foam versus ointment in patients with psoriasis vulgaris. Semin Cutan Med Surg. 2015;34 S1:PA-42.
- [Derived] Iversen L, Kurvits M, Snel-Prento AM, Menter A. Calcipotriol/Betamethasone Dipropionate Cutaneous Foam Treatment for Psoriasis in Patients With BSA 5-15% and PGA >/= 3: Post-Hoc Analysis From Three Randomized Controlled Trials. Dermatol Ther (Heidelb). 2020 Oct;10(5):1111-1120. doi: 10.1007/s13555-020-00419-2. Epub 2020 Aug 12. PMID 32785881
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 10-May-2012 Last Subject Last Visit: 19-Sep-2012
Pre-assignment Details: Prior to random., the subjects entered a washout phase (if required) where antipsoriatic treatm. and other relevant medication/treatms. had to be discontinued as defined by the excl. criteria. Depending on prior use of disallowed treatms, the washout/screening phase could last for up to 4 w prior to the first admin. of investigational products.
Groups:
- Calcipotriol Plus BDP Ointment: Calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate) ointment
- LEO 90100 Vehicle: Aerosol foam with no active ingredients
Period: Overall Study
Arm/Group | LEO 90100 | Calcipotriol Plus BDP Ointment | LEO 90100 Vehicle | Ointment Vehicle
Started | 141 | 135 | 49 | 51
Completed | 136 | 127 | 47 | 48
Not Completed | 5 | 8 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 90100 | Calcipotriol Plus BDP Ointment | LEO 90100 Vehicle | Ointment Vehicle | Total
Number analyzed (Participants) | 141 | 135 | 49 | 51 | 376
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (12.9) | 50.6 (13.1) | 45.8 (13.7) | 52.6 (11.1) | 50.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 48 | 19 | 21 | 142
  Male | 87 | 87 | 30 | 30 | 234

OUTCOME MEASURES:

1. Primary Outcome: Subjects With 'Controlled Disease' ('Clear'/'Almost Clear' for Subjects w. at Least Moderate Disease at Baseline, 'Clear' for Subjects With Mild Disease at Baseline) According to the Investigator's Global Assessment (IGA) on the Trunk and Limbs at Week 4.
Description: Assessment of disease severity (Plaque thickening, Scaling and Erythema) using a 5-point scale (Clear, Almost clear, Mild, Moderate, Severe), based on the condition of the disease at the time of evaluation.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | LEO 90100 | Calcipotriol Plus BDP Ointment | LEO 90100 Vehicle | Ointment Vehicle
Number analyzed (Participants) | 141 | 135 | 49 | 51
participants | 77 | 58 | 3 | 4

ADVERSE EVENTS:
Description: A total of 135 patients were randomized to the "Calcipotriol Plus BDP Ointment" study arm. However, one of the subjects returned all study medication unopened and therefore the safety analysis included only the 134 subjects that used the study medication.
Arm/Group | LEO 90100 | Calcipotriol Plus BDP Ointment | LEO 90100 Vehicle | Ointment Vehicle
Serious Adverse Events (participants affected / at risk) | 0/141 | 1/134 | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/141 | 0/134 | 0/49 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 90100 (N=141) | Calcipotriol Plus BDP Ointment (N=134) | LEO 90100 Vehicle (N=49) | Ointment Vehicle (N=51)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.